CLINICAL TRIAL: NCT02595073
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of DSXS in Patients With Moderate to Severe Atopic Dermatitis.
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone (DSXS) With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSXS 1504
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSXS topical product (Experimental): DSXS Active treatment
  Interventions: Drug: DSXS
- Placebo topical product (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSXS — Active treatment
  Other Names: Active
  Arms: DSXS topical product
Drug: Placebo — Placebo treatment
  Other Names: vehicle
  Arms: Placebo topical product

SUMMARY:
Efficacy and Safety of DSXS (Taro Pharmaceuticals, U.S.A., Inc.) in Patients with Moderate to Severe Atopic Dermatitis

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of DSXS (Taro Pharmaceuticals, U.S.A., Inc.) in Patients with Moderate to Severe Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

- male and non-pregnant females, age 6 months or older, with a confirmed diagnosis of moderate to severe atopic dermatitis (AD)

Exclusion Criteria:

- Lacks stable diagnosis of atopic dermatitis or has been diagnosed with mild atopic dermatitis.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS Topical Product: Desoximetasone (DSXS) Active treatment
  DSXS: Active treatment
Period: Overall Study
Arm/Group | DSXS Topical Product | Placebo Topical Product
Started | 61 | 63
Completed | 59 | 62
Not Completed | 2 | 1
Not completed — Progressive Disease | 0 | 1
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS Topical Product | Placebo Topical Product | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (18.8) | 41.7 (18.5) | 42.6 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 25 | 31 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 31 | 56
  Not Hispanic or Latino | 36 | 32 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 46 | 53 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Baseline Total Body Surface Area (BSA) [Mean (Standard Deviation); unit: meters squared] | 1.8 (0.2) | 1.9 (0.3) | 1.9 (0.3)
%BSA Affected with Atopic Dermatitis (AD) [Mean (Standard Deviation); unit: percent] | 23.4 (7.5) | 23.3 (10.1) | 23.4 (8.9)
Baseline Investigator Global Assessment (IGA) Score [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Almost Clear | 0 | 0 | 0
  Mild Disease | 0 | 0 | 0
  Moderate Disease | 53 | 56 | 109
  Severe Disease | 8 | 7 | 15
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI is a composite score based on the severity of four different signs of atopic dermatitis (Erythema, Induration/Papulation/Edema, Lichenification, and Excoriation rated 0 to 3 in severity) in four different areas of the body (Head/Neck, Upper Limbs, Trunk, Lower Limbs) multiplied by the percent of that specific body area affected multiplied by a weighting factor. The minimum score would be 0 and the maximum score would be 72. To be eligible for participation in this study a patient must have an EASI of at least 15 at baseline. A higher EASI value represents a more severe case of eczema.
  units on a scale | 18.8 (4.4) | 18.6 (3.6) | 18.7 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in Each Treatment Group That Have Clinical Success
Description: Clinical Success defined using the following scores at Visit 4 (Day 28 ± 2): At least a 2-grade improvement from the baseline IGA score (i.e., clear [0] or almost clear [1]) AND A score of clear or mild (0 or 1) for both erythema and induration/papulation/edema
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical Product | Placebo Topical Product
Number analyzed (Participants) | 61 | 63
Participants | 21 | 27
Statistical Analysis 1: Comparison: DSXS Topical Product vs Placebo Topical Product; Test type: Superiority; p = 0.3353, z-test, 2-tailed

2. Secondary Outcome: Change From Baseline in %BSA Affected at Day 28 ± 2
Description: The change in %BSA Affected from Visit 1 Baseline (Day 1) to Visit 4 End of Treatment (Day 28 ± 2)
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: percentage of BSA
Arm/Group | DSXS Topical Product | Placebo Topical Product
Number analyzed (Participants) | 61 | 63
percentage of BSA | -13.81 (0.99) | -13.24 (0.96)
Statistical Analysis 1: Comparison: DSXS Topical Product vs Placebo Topical Product; Test type: Superiority; p = 0.6190, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | DSXS Topical Product | Placebo Topical Product
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63
Other Adverse Events (participants affected / at risk) | 8/61 | 13/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS Topical Product (N=61) | Placebo Topical Product (N=63)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 1 (1)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Spider vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes